CLINICAL TRIAL: NCT02812121
Title: Umbilical Cord Blood Derived Mesenchymal Stem Cells Infusion for HBV-Related Acute-on-Chronic Liver Failure: A Randomized Controlled Trial
Brief Title: UC-MSC Infusion for HBV-Related Acute-on-Chronic Liver Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Bingliang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCBMSC; LBingliang (Registry Identifier: Bing-liang Lin)
Record Dates: First submitted 2016-05-27; First posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Liver Failure
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group MSC-1 (Experimental): Patients in Group MSC-1 received standard medical treatment and infusions of umbilical cord blood mesenchymal stem cells via peripheral veins once a week for 8 weeks.
  Interventions: Drug: umbilical cord blood mesenchymal stem cells
- Group MSC-2 (Experimental): Patients in Group MSC-1 received standard medical treatment and infusions of umbilical cord blood mesenchymal stem cells via peripheral veins once a week for 4 weeks.
  Interventions: Drug: umbilical cord blood mesenchymal stem cells
- Group Control (No Intervention): Patients in Group Control received standard medical treatment, including bed rest, nutritional supplementation, administration of human serum albumin (10g per day until serum albumin was 35g/L) and plasma (200 ml to 400 ml per day until the international normalized ratio was less than 1.5), anti-viral therapy, glycyrrhizin,S-adenosylmethionine and appropriate treatment for complications (such as infection, encephalopathy, hepatorenal syndrome and intestinal paralysis).

INTERVENTIONS:
Drug: umbilical cord blood mesenchymal stem cells
  Arms: Group MSC-1; Group MSC-2

SUMMARY:
Hepatitis B virus (HBV)-related acute-on-chronic liver failure (ACLF) is a severe disease with high mortality. Our previous study have demonstrated that peripheral infusion of bone marrow-derived mesenchymal stromal cells (MSCs) weekly for 4 times is safe and improves 24 weeks survival rate of ACLF patients. In this study, we intend to assess the safety and efficacy of umbilical cord blood derived MSCs for HBV-related ACLF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ACLF-which is characterized by acute hepatic insult manifesting as jaundice (serum total bilirubin ≥ 10×ULN umol/L) and coagulopathy (international normalized ratio≥ 1.5 or prothrombin activity < 40%), complicated within 4 weeks by ascites and/or encephalopathy as determined by physical examination, in patients with previously diagnosed or undiagnosed chronic liver disease;
2. Positive serum hepatitis B surface antigen (HBsAg) for more than 6 months;
3. End-stage liver disease scores ranging from 17-30,; 4.18-65 years of age.

Exclusion Criteria:

1. Serious complications within the previous 2 months (e.g. gastrointestinal bleeding, serious infection );
2. Concomitant autoimmune disease;
3. Superinfection with other hepatitis viruses;
4. Important organ dysfunctions not due to liver disease or malignancies;
5. Pregnancy and lactation;
6. Liver tumor or nodules secondary to cirrhosis proven by ultrasound, computerized tomography (CT), or magnetic resonance (MR) imaging;
7. Bioartificial liver support therapy;
8. Previous liver transplantation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse reactions after umbilical cord blood derived mesenchymal stem cells (UC-MSC) infusions. | 52 weeks
The survival time of patients after UC-MSC infusions. | 52 weeks

SECONDARY OUTCOMES:
The influence on levels of ALT (U/L) and AST (U/L) after UC-MSC infusions | 1,2,3,4,8,12,24,36,52weeks
The influence on levels of ALB(g/L) after UC-MSC infusions | 1,2,3,4,8,12,24,36,52weeks
The influence on levels of TBil (umol/L) after UC-MSC infusions | 1,2,3,4,8,12,24,36,52weeks
The influence on levels of INR after UC-MSC infusions | 1,2,3,4,8,12,24,36,52weeks
The influence on levels of MELD score, SOFA score and CTP score after UC-MSC infusions | 1,2,3,4,8,12,24,36,52weeks
The incidence of fatal complications after UC-MSC infusions. | 52 weeks
Comparison of levels of NKG2A among the groups after UC-MSC infusions | 2,4,8,12,24,36,52 weeks
Comparison of levels of NKG2D among the groups after UC-MSC infusions | 2,4,8,12,24,36,52 weeks
Comparison of levels of NKP46 among the groups after UC-MSC infusions | 2,4,8,12,24,36,52 weeks
Comparison of levels of KIR2DL1 among the groups after UC-MSC infusions | 2,4,8,12,24,36,52 weeks
Comparison of levels of KIR2DL3 among the groups after UC-MSC infusions | 2,4,8,12,24,36,52 weeks
Comparison of levels of KIR3DL1 among the groups after UC-MSC infusions | 2,4,8,12,24,36,52 weeks
Comparison of levels of perforin among the groups after UC-MSC infusions | 2,4,8,12,24,36,52 weeks
Comparison of levels of FasL among the groups after UC-MSC infusions | 2,4,8,12,24,36,52 weeks
Comparison of levels of gramzymeB among the groups after UC-MSC infusions | 2,4,8,12,24,36,52 weeks

IPD SHARING:
Plan to Share IPD: Undecided